CLINICAL TRIAL: NCT07243938
Title: A Prospective, Multi-cohort Clinical Study to Explore the Preliminary Efficacy and Safety of Zanidatamab in Combination With Tislelizumab for HER2-Positive GI Tumors: the UNION-HER2-BASKET Study
Brief Title: Phase II Basket Trial: Zanidatamab Plus Tislelizumab in HER2-Positive GI Tumors (UNION-HER2-BASKET)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNION-HER2-BASKET
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Rectal Cancer (LARC); Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma; Metastatic Colorectal Cancer (mCRC); Neoadjuvant Therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — zanidatamab; Capecitabine; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Locally Advanced Rectal Cancer Cohort (Experimental): All patients receive short-course radiotherapy (SCRT) (dose: 25 Gy, 5 Gy × 5 fractions), followed sequentially by 6 cycles of CAPOX chemotherapy combined with zanidatamab and tislelizumab. Following completion of the above treatment, patients underwent clinical complete response (cCR) assessment. Those assessed as cCR were placed on watchful waiting, while those assessed as non-cCR underwent Total Mesorectal Excision (TME). Postoperatively, investigators selected treatment regimens based on patient status.
  Interventions: Radiation: short-course radiotherapy; Drug: Zanidatamab; Drug: Tisleizumab(BGB-A317); Drug: Capecitabine; Drug: Oxaliplatin; Procedure: TME surgery
- Locally Advanced Gastric/Gastroesophageal Junction Cancer Cohort (Experimental): Subjects receive 3 cycles of zanidatamab and tislelizumab combined with SOX therapy. Following treatment completion, undergo D2 gastrectomy. Postoperatively, continue with 5 cycles of zanidatamab and tislelizumab combined with SOX adjuvant therapy.
  Interventions: Drug: Zanidatamab; Drug: Tisleizumab(BGB-A317); Drug: Oxaliplatin; Drug: S-1; Procedure: D2
- Advanced colorectal cancer cohort (Experimental): Subjects receive zanidatamab until disease progression or intolerable toxicity. Under specific circumstances, subjects may continue treatment after radiographic progression if the investigator assesses ongoing benefit; this decision will be made at the investigator's discretion.
  Interventions: Drug: Zanidatamab

INTERVENTIONS:
Radiation: short-course radiotherapy — 25Gy, 5Gy×5
  Arms: Locally Advanced Rectal Cancer Cohort
Drug: Zanidatamab — 1800mg(<70kg)/2400mg(≥70kg), IV，D1，Q3W
Drug: Tisleizumab(BGB-A317) — 200 mg，IV，D1，Q3W
  Arms: Locally Advanced Gastric/Gastroesophageal Junction Cancer Cohort; Locally Advanced Rectal Cancer Cohort
Drug: Capecitabine — 1000mg/m2/time，BID，PO，D1-14, Q3W
  Arms: Locally Advanced Rectal Cancer Cohort
Drug: Oxaliplatin — 130 mg/m2/次，IV，D1, Q3W
  Arms: Locally Advanced Gastric/Gastroesophageal Junction Cancer Cohort; Locally Advanced Rectal Cancer Cohort
Procedure: TME surgery — The surgery was performed 4 - 6 weeks after the end of neoadjuvant therapy in patients who assessed as non-cCR.
  Arms: Locally Advanced Rectal Cancer Cohort
Drug: S-1 — 40~60mg bid，po, d1~14，Q3W （S-1：BSA <1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2,50mg bid, BSA>1.5m2, 60mg bid）
  Arms: Locally Advanced Gastric/Gastroesophageal Junction Cancer Cohort
Procedure: D2 — Radical gastrectomy with D2 lymph node dissection was performed within 4-6 weeks after the completion of neoadjuvant therapy in patients without tumor progression on preoperative imaging assessment.
  Arms: Locally Advanced Gastric/Gastroesophageal Junction Cancer Cohort

SUMMARY:
This study is a prospective, multi-cohort clinical trial designed to evaluate the preliminary efficacy and safety of zanidatamab in combination with tislelizumab and chemotherapy/radiotherapy for patients with HER2-positive locally advanced or metastatic gastrointestinal tumors.

DETAILED DESCRIPTION:
This study is a prospective, multi-cohort clinical trial designed to explore the preliminary efficacy and safety of zanidatamab combined with tislelizumab and chemoradiotherapy in patients with HER2-positive locally advanced or metastatic gastrointestinal tumors. The study comprises three cohorts: ①Locally Advanced Rectal Cancer Cohort: Evaluate the preliminary efficacy of zanidatamab combined with tislelizumab and chemoradiotherapy for neoadjuvant and organ-preserving therapy in patients with HER2-positive locally advanced rectal cancer, as measured by investigator-assessed complete response rate (CR rate).②Locally Advanced Gastric/Gastroesophageal Junction Cancer Cohort:Evaluate the preliminary efficacy of zanidatamab combined with tislelizumab and chemotherapy for neoadjuvant treatment in patients with HER2-positive locally advanced gastric/gastroesophageal junction cancer based on investigator-assessed pathological complete response rate (pCR rate).③Advanced-line colorectal cancer cohort: Evaluate the preliminary efficacy of zanidatamab combined with tislelizumab in patients with HER2-positive advanced-line colorectal cancer based on investigator-assessed progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastric cancer and colorectal cancer
* Aged 18 to 75 years:
* Able to sign a written informed consent form and understand and comply with the requirements and evaluation schedule of this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* HER2-Positive: Immunohistochemistry (IHC) 3+ or IHC 2+ with FISH+ or NGS testing for high expression
* Locally advanced rectal cancer cohort:

  1. Histopathologically confirmed rectal adenocarcinoma
  2. Tumor tissue confirmed by immunohistochemistry (IHC) as pMMR (high expression of MLH1, MSH2, MSH6, and PMS2 proteins), or confirmed by PCR or NGS as MSI-L or MSS
  3. Tumor lower margin ≤10 cm from anal margin confirmed by colonoscopy, digital rectal examination, or MRI
  4. Clinical stage cT3-4N0M0/cTanyN+M0 (TNM staging per UICC/AJCC 8th edition; T and N stages assessed by MRI)
  5. Patients with one or more risk factors identified by MRI assessment: T4, tumor involvement of the mesorectal fascia (high MRF expression), extramural vascular invasion (high EMVI expression), ≥4 regional lymph node metastases (cN2), high lateral lymph node expression, or tumor margin ≤5 cm from the anal verge with strong organ preservation intent
  6. No prior antitumor therapy for rectal cancer (including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.; excludes traditional Chinese medicine/formulated Chinese medicine treatment)
* Locally Advanced Gastric/Gastroesophageal Junction Cancer Cohort:

  1. Histopathologically confirmed adenocarcinoma of the stomach or gastroesophageal junction
  2. Clinical stage III-IVa (i.e., TNM staging T3~4aN+M0 or T4bNanyM0, refer to UICC/AJCC 8th edition)
  3. No prior antitumor therapy for gastric or gastroesophageal junction adenocarcinoma (including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.; excludes traditional Chinese medicine/Chinese patent medicine treatment)
* Advanced colorectal cancer cohort:

  1. Histopathologically confirmed advanced colorectal cancer
  2. Previous systemic anticancer therapy for metastatic colorectal cancer with documented failure, including fluoropyrimidine, oxaliplatin, irinotecan, cetuximab, or bevacizumab (excluding contraindications). Prior anti-HER2 therapy permitted
  3. At least one measurable lesion defined according to RECIST 1.1
  4. Expected survival > 3 months
* Good organ function within ≤7 days prior to first study drug administration, as demonstrated by the following laboratory values:

  1. No blood or platelet transfusions or growth factor support therapy within ≤14 days prior to blood sample collection during the screening period, and must meet:
  2. ANC ≥ 1.5 x 10⁹/L
  3. Platelet count ≥ 100 x 10⁹/L
  4. Hemoglobin ≥ 90 g/L
  5. Serum creatinine ≤ 1.5 times the upper limit of normal (ULN)
  6. AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver metastases)
  7. Serum total bilirubin ≤ 1.5 times ULN (≤ 3 times ULN for patients with liver metastases)
  8. International Normalized Ratio (INR) ≤ 1.5 or Prothrombin Time ≤ 1.5 times ULN
  9. Activated partial thromboplastin time (aPTT) ≤ 1.5 times ULN
  10. Serum albumin ≥ 30 g/L
* Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to the first dose and must be willing to use highly effective contraception during the trial and for 120 days after the last dose. Male subjects with partners of childbearing potential must be surgically sterilized or agree to use highly effective contraception during the trial and for 120 days after the last dose.

Exclusion Criteria:

Subjects with any of the following conditions are ineligible for inclusion in this study:

* History of or concurrent other malignancies, except for basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or carcinoma in situ, provided complete remission was achieved at least 5 years prior to screening and no additional treatment is required or anticipated during the study period.
* Any of the following cardiovascular criteria:

  1. Cardiac chest pain occurring ≤28 days prior to the first study drug administration, defined as moderate pain limiting daily activities or exercise
  2. Symptomatic pulmonary embolism within ≤28 days prior to the first dose of study drug
  3. History of any acute myocardial infarction within ≤6 months prior to the first dose of study drug
  4. History of any New York Heart Association (NYHA) Class III or IV heart failure within ≤6 months prior to the first dose of study drug
  5. Any ventricular arrhythmia event of severity ≥ Grade 2 within ≤ 6 months prior to the first dose of the study drug
  6. History of any cerebrovascular accident within ≤6 months prior to the first dose of the study drug
  7. Corrected QT interval (QTc) (corrected using Fridericia's formula) ≥ 470 msec in females or ≥ 450 msec in males

  i) Note: If any patient's initial ECG shows a QTc interval > 450 msec (male) or > 470 msec (female), a follow-up ECG will be performed to verify the result h) Left ventricular ejection fraction (LVEF) ≤50% as assessed by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO). Follow-up assessment must use the same modality as the baseline assessment
* Any syncope or seizure occurring ≤28 days prior to the first study drug administration.
* Active autoimmune disease requiring systemic treatment within the past 2 years.
* Known history of human immunodeficiency virus (HIV) infection
* Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers (HBV DNA > 500 IU/mL) or active HCV carriers with detectable HCV RNA; Note: Inactive hepatitis B surface antigen (HBsAg) carriers and treated, stable hepatitis B patients (HBV DNA < 500 IU/mL) are eligible for enrollment
* History of interstitial lung disease, non-infectious pneumonia, or uncontrolled pulmonary conditions, including pulmonary fibrosis, acute pulmonary disease, etc.
* Severe chronic or active infections (including tuberculosis) requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to the first study drug dose. Note: Antiviral therapy is permitted for patients with viral hepatitis.
* Any condition requiring systemic treatment with corticosteroids (prednisone or equivalent >10 mg/day) or other immunosuppressive agents within ≤14 days prior to the first dose of study drug
* Hypersensitivity to any component of tislelizumab, zanidatamab，capecitabine, S-1, oxaliplatin, or any component of the container
* Any major surgery requiring general anesthesia within ≤28 days prior to the first dose of study drug
* Bleeding, thrombotic disorders, or use of anticoagulants (e.g., warfarin) or similar agents requiring therapeutic INR monitoring within 6 months prior to the first dose of study drug
* History of allogeneic stem cell transplantation or organ transplantation
* Live vaccine administration within ≤28 days prior to the first study drug dose. Note: Seasonal influenza vaccines, broadly classified as inactivated vaccines, are permitted. Inactivated COVID-19 vaccines are permitted. mRNA COVID-19 vaccines are not permitted. Intranasal influenza vaccines are live vaccines and are not permitted.
* Concurrent participation in another clinical study, unless it is an observational (non-interventional) study or the participant is in the follow-up period of an interventional study
* Inability to swallow tablets or diseases significantly affecting gastrointestinal function
* Pregnant or lactating women
* Other conditions deemed ineligible by the investigator.
* Locally Advanced Rectal Cancer Cohort:

  1. Previous treatment for rectal cancer, or clinical or imaging evidence of existing or potential distant metastasis
  2. Clinical or imaging evidence of intestinal obstruction, gastrointestinal perforation with bleeding, prior abdominal abscess, or recent (within 3 months) occurrence of gastrointestinal perforation, abdominal abscess, or intestinal obstruction; or investigator assessment indicating high risk of perforation or bleeding
  3. Assessed by the investigator as initially unresectable or unable to tolerate surgery
  4. Patient assessed by the investigator as having factors rendering them unsuitable for radiotherapy
  5. The patient has ≥2 concurrent colorectal cancer lesions
  6. Patient has contraindications for MRI examination
* Locally Advanced Gastric/Gastroesophageal Junction Cancer Cohort:

  1. Previous treatment for gastric/gastroesophageal junction cancer, or clinical/imaging evidence of existing or potential distant metastasis
  2. Clinical or imaging evidence of intestinal obstruction, gastrointestinal perforation, or bleeding; prior abdominal abscess; or recent (within 3 months) gastrointestinal perforation, abdominal abscess, or intestinal obstruction; or investigator assessment indicating high risk of perforation or bleeding
  3. Initial inoperability as assessed by the investigator, or inability of the patient to tolerate surgery
* Advanced colorectal cancer cohort:

  1. Patients with any prior histopathological or hematological ctDNA testing demonstrating mismatch repair gene deficiency (dMMR) or microsatellite instability (MSI-H)
  2. Presence of active leptomeningeal disease or uncontrolled brain metastases. Patients with previously treated brain metastases may be eligible if imaging shows stability, confirmed by repeat imaging demonstrating no progression for at least 4 weeks (Note: repeat imaging must occur during the study screening period).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CR Rate) | cCR rate should be assessed every 6-9 weeks following treatment initiation until completion of the 18 weeks therapy; pCR assessment in non-cCR patients following surgery (within 20 weeks after treatment initiation).
  The CR rate is defined as the sum of the pathological complete response rate (pCR rate) and the clinical complete response rate (cCR rate). To evaluate the preliminary efficacy of Zanidatamab in combination with Tislelizumab and chemoradiotherapy in neoadjuvant and organ-preserving treatment for patients with HER2-Positive locally advanced rectal cancer.
Pathological Complete Response Rate (pCR Rate) | Within 15 weeks
  Following completion of 9 weeks of neoadjuvant therapy, an assessment will be conducted after radical surgical treatment.
Progression-Free Survival (PFS) | Within 2 years
  The time interval from the start of the first treatment (date of administration of zenidatumab or tislelizumab) to the date of the subject's first progression (PD) as assessed by the investigator using RECIST version 1.1

SECONDARY OUTCOMES:
Adverse events (AEs) were graded according to the NCI CTCAE version 5·0 | an expected average of 2 years
  Adverse events and surgical safety
3-year disease-Free Survival | an expected average of 3 years
  The time from the first day of disease free (operation date) to local or distant recurrence, or the death event caused by any reason, whichever occurs first time.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, Ph.D., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: No